CLINICAL TRIAL: NCT07111741
Title: Comparison of Posterior Slab Cast With Total Contact Cast in the Management of Diabetic Foot Ulcers: a Randomized Controlled Trial
Brief Title: Comparison of Posterior Slab Cast With Total Contact Cast in the Management of Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ILS Hospital, Salt Lake (Other)
Responsible Party: Principal Investigator, Ghanshyam Goyal, Head of the Department, Diabetology & Diabetic Foot, ILS Hospital, saltlake, Kolkata, ILS Hospital, Salt Lake
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILSS/EC/0012-DFU/2022
Record Dates: First submitted 2025-07-14; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Diabetic Foot Ulcer (DFU); Offloading
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 51 patients with plantar diabetic foot ulcer (Active Comparator): Total contact cast used for offloading the ulcer
  Interventions: Device: Total contact cast
- 48 patients with plantar diabetic foot ulcer (Active Comparator): Posterior slab cast used for offloading the ulcer
  Interventions: Device: Posterior slab cast

INTERVENTIONS:
Device: Total contact cast — Arm with 51 patients was given total contact cast for offloading DFU
  Arms: 51 patients with plantar diabetic foot ulcer
Device: Posterior slab cast — Arm with 48 patients were given posterior slab cast for offloading DFU
  Arms: 48 patients with plantar diabetic foot ulcer

SUMMARY:
The goal of this clinical trial is to compare wound healing and foot related outcomes in people with plantar diabetic foot ulcer using Total contact cast (TCC) or Posterior slab cast (PSC). Ninety-nine people with neuropathic DFUs were randomized to use TCC (n=51) or PSC (n=48) together with standard of care for up to 6 months.

Researchers will compare rate of healing of ulcer at the end of 6 months, percentage reduction in the surface area, time taken to heal and patient satisfaction.

Participants will:

* Use TCC or PSC as off-loading till the ulcer heals for upto 6 months
* Visit the clinic once every 2 weeks for follow ups when inspection of the wound will be done for wound dressing, wound debridement and infection control when necessary

ELIGIBILITY:
Inclusion Criteria:

* People with diabetes
* a single neuropathic plantar DFU
* Ulcer belonging to Wagner grade 2 and 3

Exclusion Criteria:

* Persons with bilateral DFUs
* gout
* peripheral arterial disease (ABPI <0.8)
* stage 4 and 5 chronic kidney disease [estimated glomerular filtration rate (eGFR) <30 ml/min/m2]
* active Charcot arthropathy
* history of steroid intake within the past 3 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2023-01-04 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2024-04-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure in this study was healing of the ulcer at 6 months. | 6 months
  We compared the rate of healing of ulcers and time taken to heal.

SECONDARY OUTCOMES:
The secondary outcome measure was the rate of wound size reduction at 4 weeks and patient satisfaction. | 6 Months
  Healing rates will be measured by the percentage of ulcers healed or wound closure, based on clinical assessment and standardized wound measurement techniques (i.e., wound area reduction). Patient satisfaction was measured using the Likert scale 1-5 (1= very dissatisfied, 5=very satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- ILS Hoapital, Saltlake, Kolkata, Kolkata, West Bengal, India

REFERENCES:
- See also: A mouldable fibreglass backslab device as a novel approach to offload chronic plantar foot ulcers: A retrospective observational audit; First published: 21 August, 2024,https://doi.org/10.1002/jfa2.70001 — https://pubmed.ncbi.nlm.nih.gov/39169647/
- See also: Li B, Lin A, Huang J, Xie J, Liu Q, Yang C, Zhang Z. Total contact casts versus removable offloading interventions for the treatment of diabetic foot ulcers: a systematic review and meta-analysis. Front Endocrinol (Lausanne). 2023 Sep 26;14:1234761 — https://pubmed.ncbi.nlm.nih.gov/37822605/
- See also: A Comparative Study Between Total Contact Cast and Pressure-Relieving Ankle Foot Orthosis in Diabetic Neuropathic Foot Ulcers; PP Chakraborty et al; Journal of Diabetes Science and Technology 2015, Vol. 9(2) 302 -308 © 2014 — https://pubmed.ncbi.nlm.nih.gov/25452635/

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-07-31): https://cdn.clinicaltrials.gov/large-docs/41/NCT07111741/Prot_SAP_ICF_000.pdf